CLINICAL TRIAL: NCT03306719
Title: Circulating Cell-free Mitochondrial as a Novel Biomarker for Intra-amniotic Infection in Obstetrics
Brief Title: mtDNA as Novel Biomarker for Intra-amniotic Infection
Acronym: mtDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Herbert Kiss, MD, PhD, Medical University of Vienna
Other Study IDs: 1115/2017
Record Dates: First submitted 2017-10-01; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples and placental blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The intervention group will be women with premature preterm rupture of membranes (pProm), suffering from IAI
  Interventions: Biological: Blood sampling
- Control Group: Pregnant women without IAI
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Serial blood sampling

SUMMARY:
Finding a predictive biomarker for IAI could improve the clinical outcome for the mother and the neonate. The aim of this study is to quantify the copy number of circulating cell-free mitochondrial DNA in maternal serum and the placenta compared to controls.the investigators hypothesise that circulating cell-free mitochondrial DNA levels could help predict the likelihood of early inflammation in IAI. In addition, mitochondrial DNA could be a promotor triggering the pathogenesis of systemic inflammation.

DETAILED DESCRIPTION:
Background: Intra-amniotic infection (IAI) or chorioamnionitis is a common condition seen in obstetrics leading to labor abnormalities such as uterine atony, postpartum bleeding and preterm labor (Schrag et al., 2006). Further adverse effects such as perinatal death, asphyxia, sepsis, pneumonia, respiratory distress and especially neurodevelopmental delay and cerebral palsy are associated with IAI (Buhimschi et al., 2009; Holzman, Lin, Senagore, & Chung, 2007). Diagnosing IAI can be challenging due to its very heterogeneous clinical signs, which are often very insensitive for this condition. Clinical findings such as fever, tachycardia and maternal leukocytosis leave room for multiple differential diagnoses. During apoptosis (due to hypoxia, cell damage or infection) the cell membrane integrity is disturbed, releasing the cytoplasm into the blood circulation. Circulating cell-free mitochondrial DNA acts as a damage associated molecular pattern (DAMP) by activating the innate immune system leading to inflammation (Matzinger, 1994). These DAMPs are evolutionary conserved and have structural similarity to their bacterial ancestor (Zhang et al., 2010). Therefore, cell-free mitochondria can act as a potent agent triggering the immune system in an autoimmune manner as well as a biomarker for cell damage due to infection.

Objective: Finding a predictive biomarker for IAI could improve the clinical outcome for the mother and the neonate. The aim of this study is to quantify the copy number of circulating cell-free mitochondrial DNA in maternal serum and the placenta compared to controls. Investigators hypothesize that circulating cell-free mitochondrial DNA levels could help predict the likelihood of early inflammation in IAI. In addition, mitochondrial DNA could be a promotor triggering the pathogenesis of systemic inflammation.

Methods: For this study the investiagtors planned 2 groups each consisting of 30 patients. The control group are pregnant women without IAI. The intervention group will be women with premature preterm rupture of membranes (pProm), suffering from IAI (meeting the diagnostic criteria for IAI suggested by the National Institute of Child Health and Human Development Workshop). 12ml of venous blood will be drawn from a peripheral venous line in addition to routine blood tests, when the patient arrives at the ward (2 weeks before delivery). A further 12ml of venous blood will be taken from the peripheral venous line, during delivery (during delivery). In addition, 12ml of venous blood will be drawn from the placenta postpartum. In total, 36 ml of blood will be withdrawn in each patient. Circulating cell-free mitochondrial DNA will be quantified in maternal and placental serum by real time quantitative PCR and statistical analysis will be performed by non-parametric tests.

Design: Single center, prospective, observational pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 2 weeks before scheduled elective caesarian section at term (control group)
* Pregnant women in week 22+0 until week 28+0 who are admitted because of pPROM (intervention group)
* aged between 18 and 45 years
* Provide signed and dated informed consent

Exclusion Criteria:

* Women younger than 18 years
* No written consent
* Patients suffering from any autoimmune disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
mtDNA in Plasma | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kiss, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Biomarker pilot trial